CLINICAL TRIAL: NCT00178529
Title: Intervention for Stroke Survivors and Their Spousal Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Texas Woman's University (Other); Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NR035316
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Cerebrovascular Accident
Keywords: Stroke; Caregivers
MeSH Terms: conditions — Stroke | interventions — Counseling

INTERVENTIONS:
Behavioral: Psychoeducation, Counseling and Skill Training

SUMMARY:
This is an interdisciplinary, intervention study with stroke survivors and their spousal caregivers after discharge from a rehabilitation unit. It will determine whether couples receiving home visits from nurses and therapists over a 6 month period demonstrate better function and less psychological distress than couples who receive information by mail. All couples are visited every 3 months by a nurse who assesses their physical and psychosocial functioning.

DETAILED DESCRIPTION:
This 5-year randomized intervention study uses an advanced practice nurse, with the assistance of an interdisciplinary rehabilitation team, to provide education, support, skill training, counseling, and social and community linkages to stroke survivors and their spouses for 6 months post-hospital discharge. The intervention will be delivered using previously tested protocol guidelines. Stroke survivors and their spousal caregivers will be assessed to determine whether or not the intervention is successful in (1) improving function, quality of life and perceived health and decreasing depression in the stroke survivor; (2) decreasing unplanned clinic and emergency room visits, reducing rehospitalizations and admissions to nursing homes; (3) decreasing depression, burden, stress and improving the health of spousal caregivers and (4) decreasing cytokine imbalances related to the chronic stress of caregiving among spouses. Assessments will be made at baseline and at 3, 6, 9, and 12 months post-discharge on the stroke survivor and on the spousal caregiver by a nurse who is masked to the group assignment. To determine the effect of the intervention on cytokine imbalance, the researchers will: (1) generate cytokines from cell cultures (mitogen-induced and antigen specific T-cell lines) and (2) analyze culture supernatants and plasma samples for their immunoregulatory cytokine content. The laboratory technician and immunologist will be masked to the intervention group. All covariates (i.e., sociodemographic characteristics, severity of the stroke, dyadic relationships, family functioning, co-morbid health conditions, etc.) will be evaluated to determine which are significantly related to the outcomes and only those will be included in the model. Hierarchical Linear Models (HLM) will be used to model change over time for individual participants using a polynomial form. Depending on the nature of the change function, individual parameter estimates of the intercept, slope, and if necessary, curvature will be compared across groups.

ELIGIBILITY:
Inclusion Criteria:

Patient experienced a stroke within the last year Age 50 or older Going home with a spouse or committed partner Needs daily assistance Live within 50 miles fo the TMC Can be reached by telephone Able to understand English -

Exclusion Criteria:

Admitted from or being discharged to a nursing home Disability requiring total assistance Lethargic, obtunded or comatose Other significant CNS disease (ie, severe Parkinson's) Severe psychopathology Globally aphasic Other major illness that would interfere with rehabilitation (ie, advanced cancer) -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2001-07; Study Completion 2005-09

PRIMARY OUTCOMES:
Stroke survivor function
Stroke survivor and caregiver quality of life
Stroke survivor and caregiver stress
Stroke survivor and caregiver depression
Service utilization
Cytokine levels of caregivers

SECONDARY OUTCOMES:
Family coping styles
Social support system
Caregiver preparation
Marital relationship

CONTACTS AND LOCATIONS:
Overall Officials: Sharon K. Ostwald, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082